CLINICAL TRIAL: NCT01818362
Title: A Phase I Study to Determine the Safety and Immunogenicity of Vaccination Regimens Employing the Candidate Influenza Vaccines MVA-NP+M1 and ChAdOx1 NP+M1
Brief Title: A Phase I Study of Candidate Influenza Vaccines MVA-NP+M1 and ChAdOx1 NP+M1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLU005
Record Dates: First submitted 2013-03-18; First posted 2013-03-26 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Seasonal Influenza
Keywords: Influenza; T cells
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 2 (Experimental): ChAdOx1 NP+M1 2.5 x 10¹⁰vp followed by MVA NP+M1 1.5 x 10⁸pfu 52 weeks later.
  Interventions: Biological: MVA NP+M1; Biological: ChAdOx1 NP+M1
- Group 3 (Experimental): MVA NP+M1 1.5 x 10⁸pfu followed by ChAdOx1 NP+M1 2.5 x 10¹⁰vp 8 weeks later.
  Interventions: Biological: MVA NP+M1; Biological: ChAdOx1 NP+M1
- Group 4 (Experimental): MVA NP+M1 1.5 x 10⁸pfu followed by ChAdOx1 NP+M1 2.5 x 10¹⁰vp 52 weeks later.
  Interventions: Biological: MVA NP+M1; Biological: ChAdOx1 NP+M1
- Group 1 (Experimental): ChAdOx1 NP+M1 2.5 x 10¹⁰vp followed by MVA NP+M1 1.5 x 10⁸pfu 8 weeks later.
  Interventions: Biological: MVA NP+M1; Biological: ChAdOx1 NP+M1
- Group 5 (Experimental): ChAdOx1 NP+M1 2.5 x 10¹⁰vp
  Interventions: Biological: MVA NP+M1
- Group 6 (Experimental): ChAdOx1 NP+M1 2.5 x 10¹⁰vp followed by MVA NP+M1 1.5 x 10⁸pfu 8 weeks later.
  Interventions: Biological: MVA NP+M1; Biological: ChAdOx1 NP+M1

INTERVENTIONS:
Biological: MVA NP+M1 — MVA NP+M1 1.5 x 10⁸pfu intramuscularly.
Biological: ChAdOx1 NP+M1 — ChAdOx1 NP+M1 2.5 x 10¹⁰vp intramuscularly.
  Arms: Group 1; Group 2; Group 3; Group 4; Group 6

SUMMARY:
This will be a randomised observational phase 1 study in 48 healthy volunteers aged 18-50. The study is assessing safety and immunogenicity of viral vectored vaccines ChAdOx1 NP+M1 and MVA NP+M1 in heterologous prime-boost regimens. A crossover design will allow comparison of the two vaccines. Volunteers will be divided into 4 groups (n=12 in each group). Groups will be recruited simultaneously to control for seasonal changes in influenza. This is because at certain times of year there is likely to be a higher naturally acquired T cell response to influenza than at other times due to circulating influenza virus in the community.

The study has been extended to include 2 additional groups (group 5 & 6), each containing 12 healthy adults aged 50 years or above. Group 5 will receive ChAdOx 1 NP+M1 on day 0, and group 6 will receive this with an additional boost of MVA-NP+M1 8 weeks later.

ELIGIBILITY:
Inclusion Criteria for Groups 1-4

The volunteer must satisfy all the following criteria to be eligible for the study:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females only, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day(s) of vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Exclusion Criteria for Groups 1-4

The volunteer may not enter the study if any of the following apply:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Previous receipt of any recombinant adenoviral or recombinant MVA vectored vaccine
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled/topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Any history of anaphylaxis in reaction to vaccination
* History of cancer (except basal cell carcinoma and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any chronic illness requiring on-going or awaiting hospital specialist supervision, other than minor surgical procedures and follow up of surgery over 6 months prior to screening
* Suspected or known current injecting drug or alcohol abuse (as defined by an alcohol intake of greater than 42 units every week)
* Seropositive for hepatitis B surface (HBsAg) or hepatitis C virus (antibodies to HCV)
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* Any other significant disease, disorder or finding (including blood test results), which, in the opinion of the Investigators, would either put the volunteer at risk because of participation in the study, or may influence the result of the study
* No response / confirmation from GP regarding previous medical history

Inclusion Criteria for Groups 5-6

The volunteer must satisfy all the following criteria to be eligible for the study:

* Healthy adults aged 50 or over, no upper age limit
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For women of child bearing potential only, willingness to practice continuous effective contraception (i.e. hormonal contraception, intrauterine device or barrier contraception) during the study and a negative urinary pregnancy test on the day(s) of vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Exclusion Criteria for Groups 5-6

The volunteer may not enter the study if any of the following apply:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or plans to participate during the study period
* Previous receipt of a vaccine or plans to receive any vaccinations during the study that would interfere with the interpretation of the results of the trial
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled/topical steroids including eye drops and nasal spray/intra-articular steroid injections are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine including eggs or Kathon (a biocide added to body washes, conditioners, liquid soaps, shampoos and wipes as a preservative)
* Any history of anaphylaxis in reaction to vaccination
* History of treatment for cancer within the preceding six months (except basal cell carcinoma and cervical carcinoma in situ)
* History of serious psychiatric condition
* Any chronic illness requiring on-going or awaiting hospital specialist supervision, other than minor surgical procedures and follow up of surgery over 6 months prior to screening
* Suspected or known injecting drug abuse within the last 5 years
* Alcohol abuse (as defined by an alcohol intake of greater than 42 units every week)
* Seropositive for hepatitis B surface antigen (HBsAg) or hepatitis C virus (antibodies to HCV) or HIV
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* Any other significant disease, disorder or finding (including blood test results), which, in the opinion of the Investigators, would either put the volunteer at risk because of participation in the study, or may influence the result of the study
* No response / confirmation from GP regarding previous medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
To assess the safety of prime/boost vaccination regimens employing MVA-NP+M1 and ChAdOx1 NP+M1. | Up to 78 weeks post first vaccination.
  Safety will be assessed by the nature, frequency, severity, seriousness and duration of adverse events arising during the study combined with analysis of hematology and biochemistry lab tests for abnormalities.

SECONDARY OUTCOMES:
To assess the cellular immune response generated by prime/boost vaccination regimens employing MVA-NP+M1 and ChAdOx1 NP+M1. | 78 weeks after first vaccination
  The secondary outcomes of peak immune response after first vaccination and peak immune response after second vaccination will be analysed by calculating the area under the curve of the immune response (IFN-γ SFC/ million PBMCs) for each volunteer from baseline to week 78. The mean area under the curve in the 4 groups will then be compared using an analysis of variance, or in the case of skewed data a Kruskal Wallis test. Further pairwise comparisons will be made if a significant difference is found between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V S Hill, MD, Principal Investigator — University of Oxford
Locations (3):
- United Kingdom (3):
  - Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire
  - Surrey Clinical Research Centre, University of Surrey, Guildford
  - NIHR Wellcome Trust Clinical Research Facility Southampton, Southampton